CLINICAL TRIAL: NCT02691364
Title: Different Regulation of Immune Cells in Patients With Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jelmer Prins, MD PhD, University Medical Center Groningen
Other Study IDs: 2015/612
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Preeclampsia; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Healthy women
  Interventions: Procedure: Blood withdrawal
- Preeclamptic: Pregnant women with preeclampsia
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal

SUMMARY:
Adaptation of the maternal immune system to accommodate the semi-allogeneic fetus is necessary for pregnancy success. Dysregulation of this immune adaptation is implicated in reproductive disorders as infertility, recurrent miscarriage, fetal growth restriction, and preeclampsia. The mechanisms being responsible for fetal tolerance are not known. Several T cell subsets have been implicated in fetal tolerance. The effects of preeclampsia on memory cells are not known. The main objective of this study is to analyze the effect of preeclampsia on levels of immune cells.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* written informed consent
* 18-40 years

Exclusion Criteria:

* smoking
* immune related disorders (other than preeclampsia)
* fever / illness within the last month
* infertility
* body mass index <18 or >30

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with and without preeclampsia
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Cell levels | 1 year